CLINICAL TRIAL: NCT06300567
Title: Assessment of Patients Not Concluded After Neonatal Screening of Cystic Fibrosis, CFTR-RD Misdiagnosis.
Brief Title: Assessment of Patients Not Concluded After Neonatal Screening of Cystic Fibrosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Isabelle Sermet-Gaudelus, Professor, Hôpital Necker-Enfants Malades
Other Study IDs: CFTR-RD misdiagnosis
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: CFTR-RD
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with unconcluded diagnosis for cystic fibrosis: 1. symptomatic patientscarrying 2 variants of CFTR, including at least 1 non CF causing
  2. patients not concluded at neonatal screening of Cystic Fibrosis
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — collection of data of generated by "real world" follow up

SUMMARY:
Assessment of the outcome of patients not concluded fir cystic fibrosis, either symptomatic patients or asymptomatic children detected by newborn screening for cystic fibrosis. The aim is to identify patients potentially at risk of progressing to the clinical spectrum of cystic fibrosis

DETAILED DESCRIPTION:
Among patients not concluded for the diagnosis of cystic fibrosis, some are carriers of CFTR-RD mutations, therefore at risk of progressing to a symptomatic form, and may already have a subclinical involvement that it is important to identify. Among patients who do not carry the CFTR-RD genotype, other patients may be at risk of developing symptoms, if they are carriers of an undetected variant or wrongly classified as non-pathogenic. It is important to detect them to prevent the onset of symptoms

ELIGIBILITY:
Inclusion Criteria:

patients not concluded for the diagnosis of Cystic fibrosis either because of intermediate sweat test or because extensive genetic study has identified 2 vrainats at least 1 being not CF causing

-

Exclusion Criteria:

* patients carrying 2 CF causing variants of the CFTR gene
* patients carrying only 1 or no variants of CFTR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children of adults not concluded for the diagnosis of Cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
lung Imaging | within 3 months after visit
  abnormal lung Imaging score, assessing the area of the lung with bronchiectasis, bronchial wall thickening, mucus plug and air trapping

SECONDARY OUTCOMES:
lung infection | within 2 weeks after visit
  sputum bacterial colonization (number of Colony Forming Unit) of bacteria, fungi
pancreatic function | within 2 weeks after visit
  fecal elastase in µg/g of feces

IPD SHARING:
Plan to Share IPD: No